CLINICAL TRIAL: NCT01233362
Title: A Randomized Controlled Trial To Evaluate the Immunogenicity of Two Doses of the Modified Killed Whole-Cell Oral Cholera Vaccine Under Two Alternative Vaccination Schedules.
Brief Title: Study of Alternative Vaccination Schedule of Oral Cholera Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: National Institute of Cholera and Enteric Diseases, India (Other); Indian Council of Medical Research (Other Government); Shantha Biotechnics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR-WC-05
Record Dates: First submitted 2010-10-11; First posted 2010-11-03 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2012-08

CONDITIONS: Cholera; Diarrhoea; Vibrio Infection
Keywords: Cholera; Vaccine; Kolkata; West Bengal; India; Immunogenicity; Vaccination Schedules
MeSH Terms: conditions — Cholera; Diarrhea; Vibrio Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1: Adults; 14 days interval (Active Comparator): 89 Adults (=> 18 years aged) receiving study agents (Vaccine/Placebo) at 14 days inter-dose interval
  Interventions: Biological: Modified killed oral cholera vaccine at 14 day interval
- Arm 2: Adults; 28 days interval (Active Comparator): 89 Adults (=> 18 years aged) receiving study agents (Vaccine/Placebo) at 28 days inter-dose interval
  Interventions: Biological: Modified killed oral cholera vaccine at 28 day interval
- Arm 3: children; 14 days interval (Active Comparator): 89 children (1-17 years aged) receiving study agents (Vaccine/Placebo) at 14 days inter-dose interval
  Interventions: Biological: Modified killed oral cholera vaccine at 14 day interval
- Arm 4: children; 28 days interval (Active Comparator): 89 children (1-17 years aged) receiving study agents (Vaccine/Placebo) at 28 days inter-dose interval
  Interventions: Biological: Modified killed oral cholera vaccine at 28 day interval
- Arm 5: Adults; 14 days Interval (Active Comparator): 15 Adults (=> 18 years aged) receiving study agents (Vaccine/Placebo) at 14 days inter-dose interval
  Interventions: Biological: Modified killed oral cholera vaccine at 14 day interval
- Arm 6: Adults; 28 days interval (Active Comparator): 15 Adults (=> 18 years aged) receiving study agents (Vaccine/Placebo) at 28 days inter-dose interval
  Interventions: Biological: Modified killed oral cholera vaccine at 28 day interval

INTERVENTIONS:
Biological: Modified killed oral cholera vaccine at 14 day interval — The modified killed bivalent (O1 and O139)whole cell based oral cholera vaccine is administered orally in 2 liquid doses (without need of any buffer solution) 14 days for individuals aged 1 year and above.
  Other Names: Shancol
  Arms: Arm 1: Adults; 14 days interval; Arm 3: children; 14 days interval; Arm 5: Adults; 14 days Interval
Biological: Modified killed oral cholera vaccine at 28 day interval — The modified killed bivalent (O1 and O139)whole cell based oral cholera vaccine is administered orally in 2 liquid doses (without need of any buffer solution) 28 days for individuals aged 1 year and above; as an alternate schedule.
  Other Names: Shancol
  Arms: Arm 2: Adults; 28 days interval; Arm 4: children; 28 days interval; Arm 6: Adults; 28 days interval

SUMMARY:
The absence of a boosting response after a 14 day interval with the two-dose regimen of the modified killed oral cholera vaccine raises the possibility that a longer dosing interval may be required to observe a boost in the immune response. This study will compare the immune responses following 14-day and 28-day dosing intervals.

DETAILED DESCRIPTION:
Cholera is a re-emerging infectious disease that causes significant morbidity and mortality in populations lacking access to safe drinking water and sanitation. Provision of safe drinking water and food, establishment of adequate sanitation, and implementation of personal and community hygiene constitute the main public health interventions against cholera. These measures cannot be implemented fully in the near future in most cholera-endemic areas. Improvements to water and sanitation require substantial long-term investments, commitment from the local government and often take years to implement. In the meantime, a safe, effective, and affordable vaccine would be a useful tool for cholera prevention and control.

Considerable progress has been made during the last decade in the development of new generation oral cholera vaccines against cholera. A monovalent (anti-O1) WC-rBS oral killed cholera vaccine with a B-subunit was developed by Professor Jan Holmgren in Sweden and is sold primarily as a traveler's vaccine; and is only WHO pre-qualified vaccine till date. A version of this vaccine that lacks the B subunit and is considerably less expensive to produce ("whole-cell only") and which is now bivalent (O1 and O139), has been produced and used exclusively in Vietnam, making it the first oral cholera vaccine used primarily for endemic populations.

To internationalize the use of this improved vaccine, its production technology was modified to comply with the WHO Manufacturing practices (cGMP) standards before its manufacturing technology was transferred to an Indian manufacturing company Shantha Biotechnics Limited by the International Vaccine Institute. The modified killed bivalent oral cholera vaccine has been recently licensed by the Drugs Controller General of India (DCGI) to the Shantha Biotechnics Limited and being marketed as Shancol ® after phase II and Phase III clinical trials. It is administered orally in 2 liquid doses (without need of any buffer solution) 14 days for individuals aged 1 year and above. It was found safe, effective and provided 67% protection after two years in a placebo-controlled, randomized trial in Kolkata, India.

Despite the recent licensure, there are remaining questions that need to be answered that would be vital in deploying the vaccine including optimization of dosing regimen. A previous study performed in Kolkata revealed that two doses of the vaccine when given 14 days apart did not result in higher immune response after the first dose, contrary to earlier findings with the Swedish vaccine. This new finding may be due to the higher lipopolysaccharide (LPS) content of the modified vaccine which may have elicited sufficient immune response that it effectively blocks subsequent antigen presentation with the second dose of the vaccine.

In order to assess if immune responses will be boosted if we prolong the interval between dosing of the modified killed oral cholera vaccine, a Phase II double-blind, controlled, randomized trial to evaluate two different dosing interval schedules for the two-dose regimen will be conducted. This study will compare the immune responses following 14-day and 28-day dosing intervals. In addition to the 356 subjects for the main study, 30 subjects will be enrolled to explore the possibility of any other immunological marker for vibrio cholera infection.

ELIGIBILITY:
Healthy, non-pregnant adults aged 18 years and above and healthy children aged 1 - 17 will be recruited in Kolkata.

Inclusion Criteria:

* Males or non-pregnant females aged 18 years and above and children aged 1 -17 years who the investigator believes will comply with the requirements of the protocol (i.e. available for follow-up visits and specimen collection).
* Written informed consent obtained from the subjects or their parents/guardians, and written assent for children aged 12 - 17 years.
* Healthy subjects as determined by:

  * Medical history
  * Physical examination
  * Clinical judgment of the investigator

Exclusion Criteria:

* Ongoing serious chronic disease
* For females of reproductive age: Pregnancy (or females planning to become pregnant during the study period; as determined by verbal screening)
* Immunocompromising condition or therapy (for corticosteroids this would mean ≥0.5 mg/kg/day)
* Diarrhea (3 or more loose/watery stools within a 24-hour period) 6 weeks prior to enrollment
* One or two episodes of diarrhea lasting for more than 2 weeks in the past 6 months
* One or two episodes of abdominal pain lasting for more than 2 weeks in the past 6 months
* Intake of any anti-diarrhea medicine in the past week
* Abdominal pain or cramps, loss of appetite, nausea, general ill-feeling or vomiting in the past 24 hours
* Acute disease one week prior to enrollment, with or without fever. Temperature ≥38ºC warrants deferral of the vaccination pending recovery of the subject
* Receipt of immunoglobulin or any blood product during the past 3 months
* Receipt of antibiotics in past 14 days
* Receipt of live or killed enteric vaccine in past 4 weeks
* Receipt of killed oral cholera vaccine

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2010-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies, relative to baseline, 14 days after last dose of study agent in each dose-interval group | 14 days after the last dose of the study agent

SECONDARY OUTCOMES:
Proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies, relative to baseline, 14 days after first dose of study agent | 14 days after first dose of study agent
Geometric mean serum vibriocidal titers at baseline, 14 days after each dose of the study agent, in each dose-interval group. | 14 days after each dose of study agent
Proportion of subjects given 2 doses of study agent given 14 and 28 days apart with adverse events. | upto 1.5 months after the first dose of study agent
  Adverse events include:
  1. Immediate reactions within 30 minutes after each dose
  2. Serious Adverse Events occurring throughout the trial
  3. Reactogenicity during three consecutive days following each dose:
  Headache, vomiting, nausea, abdominal pain/cramps, gas, diarrhea, fever,loss of appetite, general ill feeling
  i. Diarrhea is defined as having 3 or more loose/watery stools within a 24 hour period.
  ii. Fever is defined as having an oral or tympanic temperature of ≥38o C
Proportion of subjects given 2 doses of vaccine given 14 and 28 days apart with significant immunological responses to the alternate assays under exploration | upto 1.5 months after the first dose of study agent
  Immunological responses to:
  Responses to:
  Fecal antibody to LPS OMP micro ELISPOT LPS-specific micro ELISPOT IgA to LPS (by ELISA) ALS assay

CONTACTS AND LOCATIONS:
Overall Officials: Dipika Sur, MD, DPH, Principal Investigator — National Institute of Cholera and Enteric Diseases, Kolkata, India
Locations (1):
- National Institute of Cholera and Enteric Diseases, Kolkata, West Bengal, India